CLINICAL TRIAL: NCT00004885
Title: CPT-11 in Combination With Weekly 24 Hour Infusion 5-FU Plus Folinic Acid Relative to Weekly 24 Hour Infusion 5-FU Plus Folinic Acid Alone in Patients With Advanced Colorectal Cancer
Brief Title: Fluorouracil and Leucovorin With or Without Irinotecan in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-40986; EORTC-40986
Record Dates: First submitted 2000-03-07; First posted 2004-04-12 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether fluorouracil and leucovorin plus irinotecan is more effective than fluorouracil and leucovorin alone for colorectal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of fluorouracil and leucovorin with or without irinotecan in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy and toxicity of high-dose fluorouracil and leucovorin calcium with or without irinotecan in patients with metastatic adenocarcinoma of the colon or rectum. II. Compare progression-free survival, overall survival, response rate, and duration of response in patients treated with these 2 regimens. III. Compare quality of life of patients treated with these 2 regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms. Arm I: Patients receive leucovorin calcium IV over 2 hours followed by fluorouracil IV over 24 hours on days 1, 8, 15, 22, 29, and 36. Arm II: Patients receive irinotecan IV over 30 minutes followed by leucovorin calcium IV over 2 hours and fluorouracil IV over 24 hours on days 1, 8, 15, 22, 29, and 36. Treatment in both arms repeats every 7 weeks in the absence of disease progression or unacceptable toxicity. Patients in arm I who develop disease progression begin second-line therapy comprising irinotecan, fluorouracil, and leucovorin calcium within 2 months of progression. Patients with complete response are taken off study after receiving treatment for one year. Quality of life is assessed before beginning study, after completion of each course, at 4 weeks after completion of study, and then every 2 months until disease progression or death. Patients are followed every 2 months until disease progression or death.

PROJECTED ACCRUAL: A total of 430 patients (215 per arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic adenocarcinoma of the colon or rectum Measurable or evaluable disease outside of any prior radiation port No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.25 times upper limit of normal (ULN) (1.5 times ULN if liver metastasis present) AST and ALT no greater than 3 times ULN (5 times ULN if liver metastasis present) Renal: Creatinine no greater than 1.25 times ULN Cardiovascular: No severe cardiac disease No uncontrolled angina pectoris No myocardial infarction within the past 6 months Gastrointestinal: No unresolved bowel obstruction or subobstruction No uncontrolled Crohn's disease or ulcerative colitis No history of chronic diarrhea Other: No second malignancy except carcinoma in situ of the cervix or nonmelanomatous skin cancer No other uncontrolled severe medical condition Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for metastatic disease No prior adjuvant chemotherapy containing topoisomerase I inhibitors At least 6 months since other prior adjuvant chemotherapy Endocrine therapy: Concurrent corticosteroids allowed Radiotherapy: See Disease Characteristics Surgery: Not specified Other: At least 4 weeks since other prior investigational drugs No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 1999-07; Primary Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus-Henning Koehne, MD, Study Chair — Klinik und Poliklinik fuer Innere Medizin - Universitaet Rostock
Locations (57):
- Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- U.Z. Gasthuisberg, Leuven, Belgium
- National Cancer Institute of Egypt, Cairo, Egypt
- Institut Gustave Roussy, Villejuif, France
- Germany (49):
  - PZB - Praxenzentrum, Aachen
  - Kreiskrankenhaus Aurich, Aurich
  - Haematology-Oncology, Braunschweig
  - Humaine Klinik Dresden GmbH, Dresden
  - Medizinische Klinik I, Dresden
  - St. Johannes Hospital - Medical Klinik II, Duisburg
  - Universitaetsklinik Duesseldorf, Düsseldorf
  - Hans-Susemihl-Krankenhaus, Emden
  - Haemato-Onkol. Praxis, Essen
  - Universitaetsklinik und Strahlenklinik - Essen, Essen
  - Kliniken Essen-Mitte, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Klinikum Frankfurt (Oder), Frankfurt (Oder)
  - Klinik Fuer Innere Medizin Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Marien Hospital, Hagen
  - Allgemeines Krankenhaus Hagen, Hagen
  - Internistisch - Onkologische Gemeinschaftspraxis, Halle
  - Martin Luther Universitaet, Halle
  - Hermann-Holthusen Institute for Radiotherapy, Hamburg
  - Haematologisch-Onkologische Praxis Altona, Hamburg
  - Evangelische Krankenhaus Hamm, Hamm
  - Henriettenstiftung - Chirurgische Klinik, Hanover
  - Krankenhaus Siloah - Medizinische Klinik II, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Marienhospital/Ruhr University Bochum, Herne
  - Universitatsklinik, Saarland, Homburg/Saar
  - Haematologisch-Oncologische Praxis, Koblenz
  - Klinikum Lippe-Lemgo, Lemgo
  - Stift Bethlehem, Ludwigslust
  - Staedtisches Klinikum Magdeburg, Magdeburg
  - Otto-Von-Guericke-Universitaet Magdeburg, Magdeburg
  - Johannes Gutenberg University, Mainz
  - Muenchen Onkol. Praxis Elisenhof, Munich
  - Praxis Innere Medizin, Neustadt
  - Kreiskrankenhaus Neustadt A. Rbge. des Landkreises Hannover, Neustadt
  - Klinikum Nurnberg, Nuremberg (Nurnberg)
  - Klinikum Ernst Von Bergmann, Postdam
  - Klinikum D. Ch. Erxleben, Quedlinburg
  - Kreiskrankenhaus Riesa, Riesa
  - University of Rostock, Rostock
  - Fachkrankenhaus Marienstift, Schwarzenberg
  - Katharinenhospital, Stuttgart
  - Eberhard Karls Universitaet, Tübingen
  - Klinikum der Universitaet Ulm, Ulm
  - Harz-Klinikum Wernigerode GMBH - Medizinische Klinik, Wernigerode
  - Klinikum der Stadt Wolfsburg, Wolfsburg
  - Gemeinschaftspraxis, Worms
  - Witten University - Klinikum Wuppertal, Wuppertal
  - Medizinische Poliklinik, Universitaet Wuerzburg, Würzburg
- Ospedale San Lazzaro, Alba, Italy
- Saint Laurentius Ziekenhuis, Roermond, Netherlands
- Russian Academy of Medical Sciences Cancer Research Center, Moscow, Russia
- Medical Oncology Centre of Rosebank, Johannesburg, South Africa

REFERENCES:
- [Result] Kohne CH, van Cutsem E, Wils J, Bokemeyer C, El-Serafi M, Lutz MP, Lorenz M, Reichardt P, Ruckle-Lanz H, Frickhofen N, Fuchs R, Mergenthaler HG, Langenbuch T, Vanhoefer U, Rougier P, Voigtmann R, Muller L, Genicot B, Anak O, Nordlinger B; European Organisation for Research and Treatment of Cancer Gastrointestinal Group. Phase III study of weekly high-dose infusional fluorouracil plus folinic acid with or without irinotecan in patients with metastatic colorectal cancer: European Organisation for Research and Treatment of Cancer Gastrointestinal Group Study 40986. J Clin Oncol. 2005 Aug 1;23(22):4856-65. doi: 10.1200/JCO.2005.05.546. Epub 2005 Jun 6. PMID 15939923
- [Result] Kohne CH, Van Custem E, Wils JA, et al.: Irinotecan improves the activity of the AIO regimen in metastatic colorectal cancer: results of EORTC GI Group study 40986. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1018, 2003.
- [Result] Kohne C, van Cutsem E, Wils J, et al.: Weekly high dose infusional 5-FU plus folinic acid (FA) with or without irinotecan (IRI) in metastatic colorectal cancer (MCRC): interim safety results of EORTC study 40986. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-532, 2002.